CLINICAL TRIAL: NCT01953536
Title: A Phase IIa Open Label, Randomized Clinical Trial to Study the Safety and Efficacy of Vintafolide and the Combination of Vintafolide and Paclitaxel Compared to Paclitaxel in Subjects With Advanced Triple Negative Breast Cancer Using Etarfolatide (EC20) Subject Selection
Brief Title: Safety and Efficacy Study of Vintafolide and Vintafolide Plus Paclitaxel Compared to Paclitaxel Alone in Participants With Triple Negative Breast Cancer (TNBC) (MK-8109-004)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Endocyte (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8109-004; 2012-005170-65 (EudraCT Number)
Record Dates: First submitted 2013-09-25; First posted 2013-10-01 (Estimated); Last update posted 2014-12-19 (Estimated); Status verified 2014-12

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — EC145; Paclitaxel; technetium 99m etarfolatide; Folic Acid; Premedication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Vintafolide (Experimental): Participants receive intravenous (IV) vintafolide 2.5 mg on Days 1, 3, 5, 15, 17, and 19 of a 28-day cycle.
  Interventions: Drug: Vintafolide 2.5 mg; Drug: Etarfolatide; Drug: Folic acid
- Vintafolide + Paclitaxel (Experimental): Participants receive IV vintafolide 2.5 mg on Days 1, 3, 5, 15, 17, and 19 of one 28-day cycle and receive IV paclitaxel on Days 1, 8, 15, and 22 of a 28-day cycle.
  Interventions: Drug: Vintafolide 2.5 mg; Drug: Paclitaxel 80 mg/m^2; Drug: Etarfolatide; Drug: Folic acid; Drug: Premedication for Paclitaxel
- Paclitaxel (Active Comparator): Participants receive IV paclitaxel on Days 1, 8, 15, and 22 of a 28-day cycle.
  Interventions: Drug: Paclitaxel 80 mg/m^2; Drug: Etarfolatide; Drug: Folic acid; Drug: Premedication for Paclitaxel

INTERVENTIONS:
Drug: Vintafolide 2.5 mg — During treatment, participants receive IV vintafolide 2.5 mg.
  Arms: Vintafolide; Vintafolide + Paclitaxel
Drug: Paclitaxel 80 mg/m^2 — During treatment, participants receive IV paclitaxel 80 mg/m^2.
  Arms: Paclitaxel; Vintafolide + Paclitaxel
Drug: Etarfolatide — During screening and prior to screening CT scan, participants receive an IV injection of 0.1 mg etarfolatide radiolabeled with 20 to 25 milliCuries of technetium-99m.
Drug: Folic acid — During screening and prior to etarfolatide injection and screening CT scan, participants receive an IV injection of 0.5 mg folic acid.
Drug: Premedication for Paclitaxel — During treatment, participants receive dexamethasone 20 mg orally 12 to 6 hours prior to paclitaxel; OR promethazine 25 mg or 50 mg IV 30 to 60 minutes prior to paclitaxel; OR cimetidine 300 mg IV or ranitidine 50 mg IV 30 to 60 minutes prior to paclitaxel.
  Arms: Paclitaxel; Vintafolide + Paclitaxel

SUMMARY:
The purpose of this study is to assess the efficacy and safety of vintafolide alone compared to vintafolide plus paclitaxel and paclitaxel alone in participants with with 100% positive folate receptor (FR) triple negative breast cancer (TNBC).

The primary hypothesis of this study is the vintafolide alone and/or vintafolide + paclitaxel will improve progression free survival (PFS) in participants with FR (100%) TNBC compared to paclitaxel alone.

DETAILED DESCRIPTION:
During the screening stage, participants will be required to have a diagnostic computed tomography (CT) scan with etarfolatide (EC20) to identify target lesions and determine eligibility for treatment. After successful screening, during the treatment stage, participants will receive study drug (vintafolide, vintafolide + paclitaxel, or paclitaxel) for approximately four 28-day cycles.

ELIGIBILITY:
Inclusion Criteria:

* Female with histologically or cytologically confirmed estrogen receptor negative, progesterone receptor negative, human epidermal growth factor receptor 2 (HER-2) negative advanced breast cancer that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective.
* Has developed progressive disease following at least 1 (and not more than 4) prior chemotherapeutic regimens for breast cancer, which was administered for treatment of locally advanced, locally recurrent and/or metastatic disease. [At least 1 regimen must have included a taxane (e.g., paclitaxel, docetaxel) in any combination or order.]
* Has at least a single measurable target lesion on a radiological evaluation that is conducted no more than 4 weeks prior to beginning of study drug. (Measurable lesions should not have received prior radiation therapy.)
* Has not received chemotherapy for 4 weeks prior to the initiation of study drug and must have recovered to ≤Common Terminology Criteria for Adverse Events (CTCAE) grade 1 toxicities related to prior chemotherapies.
* Female participants of childbearing potential should have a negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of study drug.
* Female participants of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 30 days after the last dose of study drug.
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Has no history of a prior malignancy with the exception of cervical intraepithelial neoplasia; basal cell carcinoma of the skin or has undergone potentially curative therapy with no evidence of that disease for 5 years.
* Has adequate organ function.

Exclusion Criteria:

* Has had chemotherapy, radiotherapy, or biological therapy (including monoclonal antibodies) within 4 weeks prior to study drug administration or has not recovered (≤Grade 1 or baseline) from adverse experiences due to agents administered more than 4 weeks earlier.
* Is currently participating or has participated in a study with an investigational compound or device within 28 days of initial dosing on this study.
* Has received more than 4 prior cytotoxic regimens for metastatic disease. Adjuvant treatments would not count towards this criterion.
* Has a primary central nervous system (CNS) tumor.
* Has active CNS metastases and/or carcinomatous meningitis.
* Has had prior therapy with vinorelbine (Navelbine®) or vinca-containing compounds.
* Has known hypersensitivity to paclitaxel, docetaxel, other taxane therapies, drugs formulated with polyoxyethylated castor oil (Cremophor EL®), vinblastine, other vinca derived therapies, or their components or analogs.
* Has pre-existing neuropathy >Grade 2.
* Has a recent (i.e., ≤6 weeks) history of abdominal surgery or peritonitis.
* Has a bowel occlusion or sub-occlusion.
* Has had prior abdominal or pelvic radiation therapy, or radiation therapy to >10% of the bone marrow at any time in the past, or prior radiation therapy within the last 3 years to the breast/sternum, dermal lesions, head, or neck.
* Requires anti-folate therapy.
* Has known psychiatric or substance abuse disorders.
* Is a known regular user (including "recreational use") of any illicit drugs or had a recent history (within the last year) of drug or alcohol abuse.
* Is expecting to reproduce within the projected duration of the study, and women who are pregnant or breastfeeding.
* Is known to be Human Immunodeficiency Virus (HIV)-positive.
* Has known active Hepatitis B or C.
* Has symptomatic ascites or pleural effusion.
* Has had a prior stem cell or bone marrow transplant.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-04; Primary Completion 2016-11 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | Up to 60 months

SECONDARY OUTCOMES:
Objective Response Rate (Complete Response [CR] + Partial Response [PR]) | Up to 60 months
Clinical Benefit Rate (CR + PR + Stable Disease [SD] for >=6 months) | Up to 60 months
Overall Survival (OS) | Up to 60 months